CLINICAL TRIAL: NCT03395808
Title: A Phase 3, Multicenter, Single-Arm, Open-Label Study to Evaluate the Safety of Tramadol Infusion (AVE-901) in the Management of Post-Operative Pain Following Surgery
Brief Title: Evaluate Safety of Tramadol in the Management of Postoperative Pain Following Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avenue Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AVE-901-104
Record Dates: First submitted 2017-12-22; First posted 2018-01-10 (Actual); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2019-06

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AVE-901 50mg (Other): IV Tramadol
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Tramadol — IV; 50 mg given at Hours 0, 2, 4, 8 and every 4 hours thereafter, for a total of up to 43 doses

SUMMARY:
The study evaluates the safety of IV tramadol managing post-operative pain following surgery.

DETAILED DESCRIPTION:
(Non-clinical summary) Tramadol is a centrally-acting synthetic analgesic of the aminocyclohexanol group with opioidlike effects. Tramadol is extensively metabolized following administration, which results in a number of enantiomeric metabolites that display different opioid-receptor binding properties, and monoaminergic reuptake inhibition.

ELIGIBILITY:
Inclusion Criteria:

* The patient is male or female 18-75 years of age
* Willing to give consent and able to understand the study procedures
* Female patients must be of non-childbearing potential or be practicing a highly effective contraption
* The patient must be willing to be housed in a healthcare facility and able to receive parenteral analgesia for at least 24 hours after surgery
* The patient meets definition of American Society of Anesthesiologists (ASA) Physical Class 1, or 2.

Exclusion Criteria:

* The patient has used chronic opioid therapy, defined as >= 20 MEQs of morphine per day >=3 days out of 7 days over the past 4 weeks.
* The patient has a recent (within 2 years) and/or current history of alcohol, opiate or tranquilizer abuse or dependence.
* The patient is taking herbal or dietary supplements or medications that are moderate or strong inhibitors of CYP2D6 or CYP3A4 (e.g., fluoxetine, paroxetine, amitriptyline, quinidine, ketoconazole, erythromycin, grapefruit juice) or inducers of CYP3A4 (e.g., carbamazepine, rifampin, St. John's Wort) and cannot go through a minimum washout period of 7 days prior to surgery.
* The patient has a history of epilepsy, is susceptible to seizures.
* The patient cannot be withdrawn from medications (at least 7 days prior to surgery) that may lower the seizure threshold (e.g. anti-psychotic agents, MAOI inhibitors) or which increase serotonergic tone (e.g. selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, triptans, amphetamines).
* The patient has had a recent (within 6 months) cardiovascular event or clinically significant abnormal ECG finding at screening.
* The patient has a history of Long QT Syndrome or a relative with this condition.
* The patient has expressed suicidal ideation within the past 3 months or is considered to be at risk of suicide.
* The patient is morbidly obese (body mass index [BMI] ≥ 40 kg/m2) or has documented sleep apnea requiring CPAP or other treatment.
* Female patient is pregnant and/or undergoing a pregnancy-related surgery, or breastfeeding.
* The patient has a history of cardiopulmonary, neurological or psychiatric condition that may confound the assessments of efficacy or safety.
* The patient has cirrhosis, moderate or severe hepatic impairment or an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value > 3X upper limit of normal (ULN) at Screening.
* The patient has severe renal impairment or a serum creatinine value of > 2x upper limit of normal (ULN) at Screening.
* The patient has potassium, sodium, calcium or magnesium levels outside of the normal range at Screening.
* The patient has a hemoglobin level at screening which, in the judgment of the Investigator, is not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Clinical Research, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AVE-901 50mg
Started | 251
Completed | 251
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AVE-901 50mg
Number analyzed (Participants) | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 201
  >=65 years | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151
  Male | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 85
  Not Hispanic or Latino | 166
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 43
  White | 203
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 251

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Reported Adverse Events
Time Frame: Up to 21 days
Measure: Count of Participants; unit: Participants
Groups:
- IV Tramadol 50 mg: 50 mg IV tramadol given at 0, 2, 4 hours and every 4 hours after
Arm/Group | IV Tramadol 50 mg
Number analyzed (Participants) | 251
Participants | 251

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | AVE-901 50mg
All-Cause Mortality (participants affected / at risk) | 0/251
Serious Adverse Events (participants affected / at risk) | 2/251
Other Adverse Events (participants affected / at risk) | 149/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVE-901 50mg (N=251)
Post procedural hematoma (Investigations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AVE-901 50mg (N=251)
Nausea (Gastrointestinal disorders) | 72
Vomitting (Gastrointestinal disorders) | 49
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 17
Blood creatine phosphokinase increased (Investigations) | 16
Constipation (Gastrointestinal disorders) | 14
Infusion Site pain (General disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT03395808/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT03395808/SAP_001.pdf